CLINICAL TRIAL: NCT06314802
Title: Evaluation of the Learning Curve of the Shouldice Procedure
Brief Title: Learning Curve of the Shouldice Procedure
Acronym: LCSR
Status: Recruiting | Type: Observational
Sponsor: Shouldice Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LCSR
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Groin Hernia; Shouldice Procedure
Keywords: Inguinal hernia; Shouldice repair; Learning curve
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Learning curve of Surgeon I
  Interventions: Other: no intervention
- Learning curve of Surgeon II
  Interventions: Other: no intervention
- Learning curve of Surgeon III
  Interventions: Other: no intervention
- Learning curve of Surgeon IV
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — No intervention

SUMMARY:
Hernia repair surgery is common, especially the Shouldice repair for primary inguinal hernias, which is considered a top-notch nonmesh technique. However, outcomes can vary, possibly due to differences in surgical skill and experience. Many surgeons are trained more in mesh repairs like the Lichtenstein technique, rather than nonmesh repairs like Shouldice.

Understanding a surgeon's learning curve-how many surgeries they need to do to become proficient-is crucial. Yet, there's not much research on this for the Shouldice repair. This project aims to fill that gap and improve surgeon education.

The study's goal is to find out how the learning curve affects Shouldice repair for primary inguinal hernias. They'll look at how operative time changes over a surgeon's first 300 repairs compared to their 900-1000th. They'll also check for complications and recurrence rates.

The study objectives are:

1. Explore the learning curve and factors affecting Shouldice repair.
2. Compare operative times between a surgeon's early and later surgeries.
3. Look at complications during the learning curve.
4. Determine how long training takes at Shouldice Hospital and the surgeons' previous experience.
5. Review recurrence rates between the first 300 and 900-1000 surgeries.

This research aims to give surgeons and the hernia community valuable insights into improving surgical techniques and patient outcomes.

DETAILED DESCRIPTION:
Hernia repair is one of the most commonly performed general surgeries [1]. Shouldice repair for primary inguinal hernias is a well-known and documented surgical technique [2,3] and considered to be the gold standard nonmesh hernia repair [1]. The results in the literature for a Shouldice primary inguinal hernia repair vary greatly [2,4,5], and may be due to a lack of accuracy in performing the repair [5,6] and/or lack of surgical volume and experience [7-9]. An added contributing factor could be that nonmesh repairs are not principally taught to many residents, instead the primary method taught is the Lichtenstein repair [10], which leaves out early training of nonmesh repairs, like the Shouldice Repair.

Learning curve can evaluate surgeons' performance and status (trainee or expert), which is done by determining the minimum number of procedures it takes to reach similar outcomes as known expert surgeons [10]. However, there is limited research that describes learning curve and the minimum number of hernia techniques to perform before being considered proficient [1,11]. Some research has performed analysis, which focused on operating times, to determine the learning curve for the Lichtenstein [10] and similar learning and proficiency research on TAPP [12] hernia repair procedures.

The rationale for this project is to supply valuable information to general surgeon trainees and experts, as well as the broader hernia community. There is little to no research done on the learning curve of the Shouldice repair for primary inguinal hernias and the importance of offering and learning nonmesh hernia repairs are associated with the risk of complications after mesh use, as well as treating patients who would prefer a nonmesh repairs [1]. Therefore, the significance of this project is to improve the understanding and knowledge regarding Shouldice Repair and increase surgeon education.

The purpose of this study is to determine the learning curve of a Shouldice repair for primary inguinal hernias. The primary endpoint is differences in operative length while secondarily evaluating recurrence rate and other complications.

Study Objectives:

1. To examine the learning curve and contributing variables of a Shouldice primary inguinal hernia repair
2. To compare operative time between a surgeons first 300 Shouldice primary inguinal hernia repairs and their 900-1000
3. To review learning curve and postoperative complications.
4. To determine the training period at Shouldice Hospital and examine prior experience of surgeons.
5. To review mean time to recurrence during a surgeon's first 300 Shouldice primary inguinal hernia repairs and their 900-1000

The proposed project is a pilot study consisting of a retrospective review to collect information on the learning curve of a Shouldice primary inguinal hernia repair, done at Shouldice Hospital. The study will consist of surgeons who worked at Shouldice Hospital in 2023, were hired within the past 10 years, and performed a minimum of 1000 primary inguinal hernia repairs. We estimate 4 surgeons to be included. The study will compare surgeons' first 300 Shouldice primary inguinal hernia repairs to their 900-1000. The parameters of 300 and 1000 hernia repairs were chosen based on previous publications [1,3], which used those benchmarks to indicate proficiency and expertise of the repair. We will analyze the learning curve by using operating time which has also been done for Lichtenstein [10] and similar research in TAPP [12] hernia repairs.

1. The HerniaSurge Group (2018) International guidelines for groin hernia management. Hernia 22:1-165. https:// doi. org/ 10. 1007/s10029- 017- 1668-x
2. Shouldice EB (2003) The Shouldice repair for groin hernias. Surg Clin N Am 83:1163-1187
3. Mainprize, M., Spencer Netto, F.A.C., Degani, C. et al. The Shouldice Method: an expert's consensus. Hernia 27, 147-156 (2023). https://doi.org/10.1007/s10029-022-02658-y
4. Shouldice EB (2010) Surgery illustrated-surgical atlas. the Shouldice natural tissue repair for inguinal hernia. BJUI 105:428-439
5. Lorenz R, Arlt G, Fortelny R, Gorjanc J, Koch A, Morrison J,Oprea V, Campanelli G (2020) Shouldice standard 2020: review of the current literature an results of an international consensus meeting. Hernia 25(5):1199-1207
6. Malik A, Bell CM, Stukel TA, Urbach DR (2016) Recurrence of inguinal hernias repaired in a large hernia surgical speciality hospital and general hospitals in Ontario. Can J Surg 59(1):19-25
7. Andresen K, Friis-Andersen H, Rosenberg J (2016) Laparoscopic repair of primary inguinal hernia performed in public hospitals or low-volume centers have increased risk of reoperation for recurrence. Surg Innov 23:142-147
8. Kockerling F, Bitter R, Kraft B, Hukauf M, Kuthe A, Schug-Pass C (2017) Does surgeons volume matter in the outcome of endoscopic inguinal hernia repair? Surg Endosc 31:573-585
9. Nordin P, van der Linden W (2008) Volume of procedures and risk of recurrence after repair of gorin hernias: national register study. Br Med J 336:934-937
10. Merola G, Cavallaro G, Iorio O, Frascio M, Pontecorvi E, Corcione F, Andreuccetti J, Pignata G, Stabilini C, and Bracale U. Learning curve in open inguinal hernia repair: a quality improvement multicentre study about Lichtenstein technique. Hernia (2020) 24:651-659. https://doi.org/10.1007/s10029-019-02064-x
11. Simons MP, Aufenacker T, Bay-Nielsen M, Bouillot JL, Campanelli G, Conze J, de Lange D, Fortelny R, Heikkinen T, Kingsnorth A, Kukleta J, Morales-Conde S, Nordin P, Schumpelick V, Smedberg S, Smietanski M, Weber G, Miserez M. European Hernia Society guidelines on the treatment of inguinal hernia in adult patients. Hernia (2009) 13:343-403.
12. Brucchi F, Ferraina F, Masci E, Ferrara D, Bottero L, and Faillace GG. Standardization and learning curve in laparoscopic hernia repair: experience of a high-volume center. BMC Surgery (2023) 23:212. https://doi.org/10.1186/s12893-023-02119-y

Supplemental Material:

ELIGIBILITY:
Inclusion Criteria:

* A surgeon, who operated on at least 1000 primary inguinal hernias using the Shouldice technique
* Surgeon at the shouldice hospital

Exclusion Criteria:

* A surgeon, who operated on less than 1000 primary inguinal hernias using the Shouldice technique

Ages: 16 Years to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study Population:
  The study population will include male and female patients aged 16-90 years of age, standard age of patients accepted for surgery at Shouldice Hospital, who had a Shouldice repair of a primary inguinal hernia at Shouldice Hospital, all nationalities and races, capable of speaking and reading English, in good general health, and there is no geographic location constraint. Patients will be excluded if they underwent a mesh repair, repair of a scrotal hernia, non-Shouldice or modified Shouldice tissue repair, a hernia that was not an inguinal type, recurrent hernias, repairs with bowel resection, and/or and surgery was deemed an emergency.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-05-11 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Operating time I | Operating time of shouldice primary hernia repair
  Operating time of shouldice primary hernia repair after the first 300 cases

SECONDARY OUTCOMES:
Operating time II | Operating time of shouldice primary hernia repair after the 1000 cases
  Operating time of shouldice primary hernia repair after the 1000 cases
Operating time III | Operating time of shouldice primary hernia repair after the 1000 cases
  Interindividual comparison of operating time between surgeon I, II, III and IV

CONTACTS AND LOCATIONS:
Locations (1):
- Shouldice hospital, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided